CLINICAL TRIAL: NCT05654610
Title: Real-world Evidence Study on the Performance and Safety of the Medical Device Halova Ovules in the Local Treatment of Vaginal Atrophy
Brief Title: Real-world Evidence Study on the Performance and Safety of Halova Ovules
Status: Completed | Type: Observational
Sponsor: Perfect Care Distribution (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Other Study IDs: HALOVRW/01/2022
Record Dates: First submitted 2022-11-18; First posted 2022-12-16 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Vaginal Atrophy
Keywords: Dyspareunia; Dysuria; Vaginal lubrication
MeSH Terms: conditions — Dyspareunia; Dysuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Halova — Halova is a class I medical device formulated as vaginal ovules and intended for intravaginal administration in order to promote and/or accelerate the hydration, healing, re-epithelialization and/or soothing of injured, atrophic or irritated vaginal mucosa. The ovules melt evenly in the vaginal mucosa forming a cream with a moisturizing and calming effect that support the restoration of the vaginal epithelium.

SUMMARY:
An open-label, multicentric, non-randomized, single-arm, pilot, interventional clinical investigation to confirm the tolerability and performance of the medical device Halova in lubrication of the vagina and vaginal atrophy treatment.

DETAILED DESCRIPTION:
The primary objective of this investigation is to evaluate the therapeutic performance and tolerability of Halova ovules in treating vaginal atrophy and restoring the natural lubrication of the vaginal mucosa.

The secondary objective of this clinical investigation are to evaluate the performance of the medical device by clinical examination, and the degree of patient satisfaction related to the intended use (Likert scale).

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged between 18 and above, in pre-menopause or menopause;
* Adult women with atrophic vaginitis caused by estrogen hormone deficiency;
* Adult women who have vaginal dryness as a result of contraceptive treatment or other disorders;
* Subjects with a normal cervical cytology report, e.g. Negative for intraepithelial lesions or malignancy (NILM) or slightly changed to atypical squamous cells of undetermined significance (ASC-US) in the last 6 months;
* Subjects willing to provide signed informed consent for participation in clinical investigation.

Exclusion Criteria:

* Subjects with vulvar or cervical cancer.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Halova is a medical device intended for intravaginal administration.
Study Population: Adult women, with atrophic vaginitis caused by estrogen hormone deficiency or vaginal dryness as a result of contraceptive treatment or other disorders.
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Rating and assessing of treatment-related Adverse Events | 30 days
  The safety of Halova® ovules as measured by the rate of treatment-related adverse events, including serious adverse events (SAEs), in subjects participating in the clinical investigation

SECONDARY OUTCOMES:
Clinical Performance | 30 days
  Evaluation by the Investigator of the disorder-related symptoms
Patient Satisfaction | 30 days
  The degree of satisfaction when using the medical device will be assessed using a five-point Likert Scale from Very satisfied to Very unsatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Ema Peta, Study Director — Perfect Care Distribution
Locations (14):
- Romania (14):
  - Spitalul Clinic Dr. Ion Cantacuzino Bucharest, Bucharest
  - Med Life Humanitas Cluj-Napoca, Cluj-Napoca
  - Cabinet Medical - Dr. Saleh K. Majed, Craiova
  - Cabinet Medical - Dr. Surpanelu Oana, Iași
  - MediBlue, Iași
  - Clinica Natisan Pitesti, Piteşti
  - Cabinet Dr. Rădulescu G. Mihaela Elena, Râmnicu Vâlcea
  - Ramnicu Valcea, Râmnicu Vâlcea
  - Cabinet Ginecologic Dr. Popescu Sibiu, Sibiu
  - Clinica iMED, Sibiu
  - Pan Medical Sibiu, Sibiu
  - Bradmed SRL, Târgu Jiu
  - Clinica Medicala Dr. Cioata Ionel Trifon, Timișoara
  - Spitalul Judetean de Urgenta Tulcea, Tulcea